CLINICAL TRIAL: NCT05537844
Title: Longitudinal Sample Collection to Investigate Adaptation and Evolution of Ovarian High-grade Serous Carcinoma
Acronym: BriTROC-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liz-Anne Lewsley (Other)
Collaborators: Ovarian Cancer Action (Unknown)
Responsible Party: Sponsor-Investigator, Liz-Anne Lewsley, Project Manager, Cancer Research UK, Glasgow
Organization: Cancer Research UK, Glasgow (Other)
Other Study IDs: BriTROC2-2019
Record Dates: First submitted 2022-09-05; First posted 2022-09-13 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Ovarian Cancer; High Grade Serous Carcinoma; Carcinosarcoma, Ovarian; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; BRCA1 Mutation; BRCA2 Mutation
MeSH Terms: conditions — Ovarian Neoplasms; Carcinosarcoma; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Tumour tissue from diagnosis from 250 patients
  2. Whole blood samples from 250 patients
  3. Plasma blood samples from 250 patients
  4. Serum blood samples from 250 patients
  5. Ascites/pleural fluid/peritoneal washings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In BriTROC-2, up to 250 women with a confirmed diagnosis of high-grade serous/high-grade endometrioid or carcinosarcoma will be eligible for full consent (Part 2) and registration to BriTROC-2 and will be followed prospectively until first relapse. Women with presumed newly-diagnosed high-grade serous carcinoma of the ovary, fallopian tube or peritoneum can be approached for consent to Part 1 (screening consent) of BriTROC-2 prior to formal diagnosis.

The aim of this study is to acquire tumour material at diagnosis and relapse, whole blood for genomic analysis and plasma for ctDNA. This study will also isolate single cells and establish organoid cultures from ascites/peritoneal washings.

DETAILED DESCRIPTION:
BriTROC-2 is a sample collection study from women with ovarian cancer from the point of diagnosis to the time of disease relapse.

Ovarian cancer has a poor prognosis. The large majority of patients with ovarian cancer will relapse and ultimately develop fatal chemotherapy resistance. Although there is a wealth of information regarding the molecular basis of ovarian cancer at diagnosis, very little is known about the drivers of treatment resistance (both intrinsic and acquired) and the processes that are active at relapse. This research requires sequential collection of tumour material for women throughout the course of their disease.

This multicentre study will collect tumour samples, ascites (fluid within the abdomen) and blood from women with newly diagnosed ovarian cancer and follow these women through to relapse of their disease. The samples collected will be used to look at patterns within the tumour to identify those that are able to predict response to chemotherapy and outcome. Assays and models will be developed that can look at the process that are active in a tumour at time of sample acquisition. This will give clues into the mechanisms that drive treatment resistance. Ultimately this research aims to guide future treatment options for women with ovarian cancer.

Recruitment will be over 3 years and this study will be conducted at sites with expertise in managing ovarian cancer and the ability to carry out the appropriate sample collection and collect high quality clinical data.

This study is the second collaborative project within the UK to collect samples from women with ovarian cancer. The success of the first study, BriTROC-1, demonstrated the feasibility of sample collection from women with relapsed ovarian cancer. The methods and frameworks established in BriTROC-1 will be used for BriTROC-2.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 years.
2. Ability to provide written informed consent prior to participating in the trial and any trial related procedures being performed.
3. Ovarian, fallopian tube or primary peritoneal carcinoma of high-grade serous, high-grade (grade 3) endometrioid or carcinosarcoma histologies.
4. Patients with ovarian, fallopian tube or primary peritoneal carcinoma of any histological subtype in patients with known germline mutations in BRCA1 or BRCA2.
5. Willingness to comply with scheduled visits, treatment plans, laboratory tests and other trial procedures.
6. Life expectancy > 6 months.
7. No contraindication to obtaining a surgical or image-guided biopsy.
8. Patients with confirmed ovarian, fallopian tube or primary peritoneal carcinoma of high-grade serous, high-grade (grade 3) endometrioid or carcinosarcoma histologies who have consented for their tissue to be collected under a generic tissue consent (i.e. have not consented to Part 1) may be eligible for full consent following discussion with the trials team.

Exclusion Criteria:

1. Ovarian, primary peritoneal or fallopian tube cancer of low grade serous, grades 1 or 2 endometrioid or clear cell subtypes unless associated with known germline mutation in BRCA1 or BRCA2
2. Borderline/low malignant potential tumours
3. Any non-epithelial ovarian malignancy
4. Diagnosis of high-grade serous cancer made on cytology only
5. Patients who have received any prior treatment for known high-grade ovarian carcinoma
6. Other severe or uncontrolled systemic disease or evidence of any other significant disorder or lab finding that makes it undesirable for the patient to participate in the trial
7. History of physical or psychiatric disorder that would prevent informed consent and compliance with protocol
8. Pregnant or lactating women
9. Patients with any other severe concurrent disease which may increase the risk associated with trial participation
10. Any psychological, familial, sociological or geographical consideration potentially hampering compliance with the trial protocol and follow up schedule.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female patients with ovarian cancer
Study Population: In BriTROC-2, a cohort of women with presumed newly-diagnosed high-grade carcinoma of the ovary, fallopian tube or peritoneum will be recruited at the time of diagnosis and approached for consent to Part 1 (screening consent) of BriTROC-2. Up to 250 women with a confirmed diagnosis of high-grade serous/high-grade endometrioid or carcinosarcoma will be eligible for full consent (Part 2) and registration to BriTROC-2 and will be followed prospectively until first relapse. The aim of this study is to acquire tumour material at diagnosis and relapse, whole blood for genomic analysis and plasma for ctDNA. This study will also isolate single cells and establish organoid cultures from ascites/peritoneal washings.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2024-10-27 (Estimated); Study Completion 2025-04-27 (Estimated)

PRIMARY OUTCOMES:
Tumour Biopsies (to be collected from 250 patients) | Through study completion, an average of 1 year
  To obtain tumour biopsies from 250 women with newly diagnosed high-grade carcinoma of the ovary, fallopian tube or peritoneum - all those with high-grade serous carcinoma (HGSC), high-grade endometrioid carcinoma or carcinosarcoma will be eligible.

SECONDARY OUTCOMES:
Whole Blood Samples for germline DNA isolation | Baseline
  To obtain whole blood for germline DNA isolation.
Plasma Blood Samples (to be collected for storage for future analyses) | Baseline and prior to Cycles 1-3 of chemotherapy (depending on treatment this could be up to 28 days), relapse
  To obtain plasma for ctDNA at diagnosis, during first line chemotherapy, at follow up and at the time of relapse.
Ascites/Peritoneal Washings (where possible from diagnosis and relapse) | Through study completion, an average of 1 year
  To obtain ascites/washings from women at diagnosis and at the time of relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Iain McNeish, Principal Investigator — Imperial College London
Locations (11):
- United Kingdom (11):
  - Bristol Haematology & Oncology Centre, Bristol
  - Addenbrookes Hospital, Cambridge
  - Western General Hospital, Edinburgh
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - St Bartholomew's Hospital, London
  - University College London Hospital, London
  - Royal Marsden Hospital NHS Trust, London
  - Hammersmith Hospital, London
  - St Mary's Hospital, Manchester
  - The Christie Hospital NHS Trust, Manchester
  - Mount Vernon Cancer Centre, Northwood

IPD SHARING:
Plan to Share IPD: Undecided